CLINICAL TRIAL: NCT06360107
Title: RCT of a Brief Video Intervention Targeting Peer Social Inclusion to Reduce Depression-related Stigma and Increase Help-seeking Among Adolescents
Brief Title: RCT of a Brief Video Intervention Targeting Peer Inclusion to Reduce Depression-related Stigma in Adolescents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Columbia University (Other)
Responsible Party: Principal Investigator, Doron Amsalem, Assistant Professor, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 76729
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Depression; Adolescent - Emotional Problem; Stigma, Social; Help-Seeking Behavior
MeSH Terms: conditions — Depression; Social Stigma; Help-Seeking Behavior

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Peer social-inclusion enhanced social contact brief video (Experimental): Novel brief video (1-2 mins) in which an adolescent talks about feeling depressed, and the impact this has on peer relationships, getting treatment, selectively disclosing mood problems with some friends, and experiencing support from both peers and family which helped facilitate recovery from depression.
  Interventions: Other: brief video
- Generic social contact brief video (Active Comparator): Similar to existing brief videos (1-2 mins), an adolescent talks about feeling depressed, and then asking parents for help, and receiving professional treatment. This video does not make any references to peers or social support.
  Interventions: Other: brief video
- Control (Other): Brief video (1-2 mins) provides information about symptoms of depression and how to seek help with computer-generated voice, to isolate mechanisms of information from identification and emotional engagement.
  Interventions: Other: brief video

INTERVENTIONS:
Other: brief video — brief video about depression

SUMMARY:
The goal of this study is to test the efficacy of a brief video intervention emphasizing peer inclusion on depression-related stigma and stigma outcomes (e.g., help seeking attitudes, secrecy) among adolescents 14-18.

Timely identification and treatment of depression in adolescents is a public health priority. However, most youth with depression do not seek treatment, and stigma has been identified as the primary barrier to help-seeking. Experiments have found brief video-based interventions (BVIs), 1-2 minute videos similar to those viewed by youth on social media platforms, based on the principle of "social contact" with individuals affected by a stigmatized condition, effective in reducing depression-related stigma and increasing help-seeking among adolescents. However, given the extreme time constraints of these videos, optimizing the messaging is paramount. Prior research has indicated that concerns about peer social inclusion are fundamental in shaping stigma among adolescents.

In this 3-arm RCT, we will recruit adolescents aged 14-18 using an online crowdsourcing platform, to test the efficacy of a) standard BVI that addresses mental health treatment but does not address concerns about peer inclusion/exclusion, b) novel BVI focused on mental health treatment and peer inclusion, and c) control condition that provides information without social contact.

DETAILED DESCRIPTION:
Brief video-based interventions (BVIs) have been studied as a means of reducing stigma toward mental health problems and increasing help-seeking among youth. "Contact-based interventions," in which a representative of a stigmatized group shares their personal stories, have been found one of the most effective anti-stigma intervention. Effective contact-based interventions target to a specific population, account for the specific interests of that population, and credibly provide stories that highlight recovery in a plausible manner to moderately disconfirm stereotypes. BVIs package contact-based stigma interventions into a format desirable to youth-- short (1-2 minute) messages in the style of social media content. Prior RCTs have tested BVIs targeting depression-related stigma in adolescents, featuring a young person describing experiences with depressive symptoms, that improved as they sought support from parents and professionals, compared to a control video of a young person discussing family and activities with no mention of mental health. Prior BVIs have not emphasized adolescent concerns about peer rejection and identity. Since existing research emphasizes the central nature of these concerns in shaping mental health-related stigma among adolescents [4, 5], BVIs that address peer social concerns may be most effective. Thus, we hypothesize that a BVI focused on peer inclusion will have greater impact on reducing stigma and increasing help-seeking than a BVI with more general content.

We will measure three distinct domains of stigma:

1. personally held attitudes,
2. perceptions of how peers may devalue and discriminate against teens with depression, and
3. secrecy (i.e., to avoid potential negative repercussions of stigma).

ELIGIBILITY:
Inclusion Criteria:

* Self-identify as English-speaking
* US residents
* 14-18 years old

Exclusion Criteria:

* Non English speakers
* Do not reside in the US
* <14 or greater than or equal to 19 years old

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 645 (Actual)
Dates: Start 2024-12-17 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Depression Stigma Scale (modified) | immediately after viewing video
  measures personally held attitudes toward depression; modified to remove element irrelevant to teens
Ultra-brief Self-stigma of Help-Seeking | immediately after viewing video
  attitudes toward seeking professional help for mental health problem

SECONDARY OUTCOMES:
Adolescent Stigma Scale (modified) | immediately after viewing video
  subscales measuring perceived societal devaluation and secrecy coping

CONTACTS AND LOCATIONS:
Overall Officials: Doron Amsalem, MD, Principal Investigator — Columbia University
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Amsalem D, Martin A. Reducing depression-related stigma and increasing treatment seeking among adolescents: randomized controlled trial of a brief video intervention. J Child Psychol Psychiatry. 2022 Feb;63(2):210-217. doi: 10.1111/jcpp.13427. Epub 2021 Apr 6. PMID 33821507